CLINICAL TRIAL: NCT03508271
Title: Real-World Comparative Effectiveness Research Among Elderly Non-valvular Atrial Fibrillation (NVAF) Patients With Heart Failure (HF) Using Oral Anticoagulants
Brief Title: Effectiveness of Oral Anticoagulants in Elderly Patients With Non-Valvular Atrial Fibrillation and Heart Failure
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-681
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Atrial Fibrillation; Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly individuals with NVAF and HF who are taking OAC's
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
Observational study of elderly individuals diagnosed with Non-Valvular Atrial Fibrillation and Heart Failure who are beginning oral blood thinners

ELIGIBILITY:
Inclusion Criteria:

* Were age greater than or equal to 65 years as of the index date
* Had greater than or equal to 1 diagnosis of AF prior to or on the index date
* Had greater than or equal to 1 diagnosis claim of HF during the 12 months prior to or on the index date
* Had 1 or more pharmacy claim for oral blood thinners

Exclusion Criteria:

* Claims indicating diagnosis or procedure for hip/knee replacement surgery within 6 weeks prior to index date
* Pharmacy claim for warfarin, apixaban, dabigatran, edoxaban or rivaroxaban during the 12-month baseline period
* Greater than 1 oral anticoagulants prescription claim on the index date and/or with a follow-up less than 1 day
* Had medical claim indicating VTE in the 12 months prior to index date

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly individuals diagnosed with NVAF (non-valvular atrial fibrillation) and HF (heart failure) who are new initiators of DOAC's (direct oral anticoagulants)
Sampling Method: Probability Sample
Enrollment: 60000 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
Incidence of stroke/systemic embolism (SE) | Approximately 195 weeks
Incidence of major bleeding | Approximately 195 weeks

SECONDARY OUTCOMES:
Incidence of miocardial infarction (MI) | Approximately 195 weeks
Incidence of all cause mortality | Approximately 195 weeks
Incidence of all cause hospitalization | Approximately 195 weeks
Incidence of major adverse cardiac event | Approximately 195 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Ann Arbor, Michigan, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm